CLINICAL TRIAL: NCT01658280
Title: Conventional Versus Ultrasound-guided Transbronchial Needle Aspiration, Using Rapid On-site Cytological Evaluation, for the Diagnosis of Hilar/Mediastinal Enlarged Lymph Nodes: a Randomized Controlled Trial.
Brief Title: Conventional Versus Ultrasound-guided Transbronchial Needle Aspiration for the Diagnosis of Hilar/Mediastinal Lymphadenopathies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Stefano Gasparini, Professor, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PAN-001
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Mediastinal Lymphadenopathy; Hilar Lymphadenopathy; Lymphoma; Lung Neoplasms; Sarcoidosis
Keywords: transbronchial needle aspiration; ultrasound guided transbronchial needle aspiration; sensitivity; hilar/mediastinal adenopathy
MeSH Terms: conditions — Lymphoma; Lung Neoplasms; Sarcoidosis; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional TBNA + ROSE (Active Comparator): Patients allocated in this group will undergo conventional TBNA, performed in a bronchoscopy suite by the same operator under conscious sedation, using 19-G needle size. Three needle passes for each approachable station will be performed. The samples obtained will be examined on-site by experienced blinded cytopathologist.
  In case of samples obtained from conventional TBNA defined as "non diagnostic", the operator will shift to the EBUS procedure.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs
  Interventions: Device: EBUS-TBNA
- EBUS-TBNA + ROSE (Experimental): Patients allocated in the intervention group will undergo EBUS-TBNA procedure, performed in a bronchoscopy suite by the same operator under conscious sedation Three needle passes for each approachable station will be performed. The samples obtained will be examined on-site by experienced blinded cytopathologist.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs
  Interventions: Device: EBUS-TBNA

INTERVENTIONS:
Device: EBUS-TBNA — Patients allocated in the intervention group will undergo EBUS-TBNA procedure, performed in a bronchoscopy suite by the same operator under conscious sedation Three needle passes for each approachable station will be performed. The samples obtained will be examined on-site by experienced blinded cytopathologist.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs

SUMMARY:
The main purpose of the present study is to assess whether the sensitivity of Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) is superior to that of conventional TBNA in the diagnosis of hilar/mediastinal adenopathy and lung cancer staging.

DETAILED DESCRIPTION:
The role of transbronchial needle aspiration (TBNA) for the diagnosis of hilar/mediastinal adenopathy and lung cancer staging is well established. However, it is a blind procedure and its diagnostic yield seems to be related to the operator experience, as well as to the size and location of lymph nodes. In the recent years, there has been increased interest in imaging-assisted TBNA and the endobronchial ultrasound has been suggested to be feasible and to improve the diagnostic yield.

Another technique able to optimize the performance of transbronchial aspirations is the rapid on-site cytological examination (ROSE), allowing to assess the adequacy of samples collected. In this context, no comparative studies between standard TBNA and EBUS-TBNA have been performed. It is very important for clinical practice to definitively assess the possible superiority of EBUS-TBNA in terms of sensitivity, and to provide information regarding safety, procedural time and costs to define the best diagnostic strategy.

The study is focused on 252 patients who have at least one hilar/mediastinal lymph node > 1 cm on CT scan in at least one approachable lymph nodal station (except 2R and 2L) for which a diagnostic cyto-histological assessment is required for clinical purpose. Patients will be randomized 1:1 (control : intervention) by a computer-generated random-allocation system to undergo EBUS-TBNA or conventional TBNA. In case of failure of conventional TBNA, the operator will shift to EBUS procedure. Moreover,a subgroup analysis will be perform to assess the potential impact of lymphnode size and position on final results(univariate analysis).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18years;
* presence of at least one hilar/mediastinal adenopathy >1 cm on short axis assessed by contrast-enhanced CT scan in at least one approachable stations other than 2R and 2L;
* ability to give an informed consent.

Exclusion Criteria:

* presence of mediastinal adenopathy in stations 2R and 2L;
* coagulopathy or bleeding diathesis that cannot be corrected;
* severe refractory hypoxemia;
* unstable hemodynamic status;
* inability to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To compare the sensitivity of EBUS-TBNA and conventional TBNA in the diagnosis of hilar/mediastinal adenopathies | 36 months
  The sensitivity is defined as the rate of true positive diagnoses/(true positive + false negative). Sensitivity of EBUS-TBNA will be considered superior to that of conventional TBNA if it will achieve at least a value of 90%

SECONDARY OUTCOMES:
Specificity of TBNA and EBUS-TBNA | 36 months
  Specificity is defined as the rate of true negatives diagnoses /true negative + false positive
Sensitivity of EBUS-TBNA performed after the possible failure of traditional TBNA | 36 months
Number of partecipants with adverse events | 36 months
Costs related to each diagnostic strategy | 36 months
  It will be evaluated the cost related to the whole procedure, including the possible shift to EBUS-TBNA.
Procedural time | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Gasparini, Professor, Principal Investigator — Azienda Ospedaliero, Universitaria Ospedali Riuniti
Locations (1):
- Pulmonary Diseases Unit, Department of Immunoallergic and Respiratory Diseases, Azienda Ospedaliero Universitaria 'Ospedali Riuniti', Ancona, The Marches, Italy

REFERENCES:
- [Background] Herth F, Becker HD, Ernst A. Conventional vs endobronchial ultrasound-guided transbronchial needle aspiration: a randomized trial. Chest. 2004 Jan;125(1):322-5. doi: 10.1378/chest.125.1.322. PMID 14718460
- [Background] Gasparini S. It is time for this 'ROSE' to flower. Respiration. 2005 Mar-Apr;72(2):129-31. doi: 10.1159/000084041. No abstract available. PMID 15824520
- [Background] Toloza EM, Harpole L, Detterbeck F, McCrory DC. Invasive staging of non-small cell lung cancer: a review of the current evidence. Chest. 2003 Jan;123(1 Suppl):157S-166S. doi: 10.1378/chest.123.1_suppl.157s. PMID 12527575